CLINICAL TRIAL: NCT00223093
Title: A Single-Center Open-Labelled Study of the Administration of Transplant-Acceptance Inducing Cells (TAIZ) for the Induction of Donor Specific Tolerance in Renal Allograft Recipients (Cadaver Kidney)
Brief Title: TAIZ -Monocytes for the Induction of Donor Specific Tolerance in Renal Allograft Recipients (Cadaver Kidney)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 006
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2005-10-28 (Estimated); Status verified 2003-04

CONDITIONS: Renal Transplantation
Keywords: renal transplantation, TAIZ-moncytes

INTERVENTIONS:
Drug: TAIZ

SUMMARY:
Induce tolerance or reduce the amount of immunosuppression after renal transplant patient (receiving cadaver kidney)with so called TAIZ-monocytes

ELIGIBILITY:
4.3.1 Inclusion Criteria

Patients must meet all the following inclusion criteria to be considered for admission to the trial:

1. Male or female adult patients aged between 18 and 64 years (inclusive). A female of childbearing potential may be enrolled provided she:

   * has a negative pregnancy test at Screening and
   * is routinely using adequate contraception prior to and during the study and
   * agrees not to attempt to become pregnant during the study and
   * is not lactating A female of non-childbearing potential will be defined as one who has been postmenopausal for at least one year or has been surgically sterilised.
2. Patients receiving a first renal transplant.
3. Patients who fulfil the criteria to receive an allogeneic renal transplant from a cadaver (according to the Eurotransplant (ET) manual on organ allocation and the Bundesärztekammer allocation criteria).
4. Patients who, after the nature of the study and the disclosure of their data has been explained to them, have freely given Informed Consent in writing.

4.3.2 Exclusion Criteria

Patients presenting any of the following exclusion criteria must not be included in the trial:

1. Patients who have received a renal transplant.
2. Patients who have an active infection at the time of entry into the study (Screening).
3. Recipient and donor pairs who show the following incompatible CMV constellation: the donor is CMV positive and the recipient is CMV negative.
4. Patients and donor who have positive evidence of HIV or have active virus hepatitis B and C.
5. Patients with a history of alcohol and/or drug abuse.
6. Patients who are pregnant women or nursing mothers.
7. Known hypersensitivity or contraindication to one of the immunosuppressives administered during the course of the study: tacrolimus, sirolimus or steroids (prednisolone and methylprednisolone).
8. Patients with a history or present symptoms of autoimmune vasculitis.
9. Detection of >5% HLA antibodies (current values determined during the last three months).
10. Patients with a malignancy or history of malignancy.
11. Patients with renal insufficiency due to a vasculitis.
12. Recipient and donor pairs with complete HLA matching.
13. Patients whose condition requires continuous systemic steroid administration.
14. Patients who are simultaneously participating or plan to participate in any other clinical study.
15. Psychiatric or emotional problems or lack of knowledge of the German language which would invalidate the giving of Informed Consent or limit the ability of the subject to comply with study requirements.
16. Unwillingness or inability to provide Informed Consent or to participate satisfactorily for the entire trial period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2004-02; Study Completion 2005-08

PRIMARY OUTCOMES:
graft survival
replacement of immunosuppressives after treatment with Transplant-Acceptance Inducing Cells (TAIC)
serum creatinine
rejection episodes
re-introduction of immunosuppressives.

SECONDARY OUTCOMES:
safety and tolerability of the treatment with Transplant-Acceptance Inducing Cells (TAIC) Adverse Events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kunzendorf, MD, Principal Investigator — University of Schleswig-Holstein, Campus Kiel Department of Nephrolgy